CLINICAL TRIAL: NCT03769844
Title: GM-CSF for Reversal of immunopAralysis in pediatriC sEpsis-induced MODS (GRACE)
Brief Title: GM-CSF for Reversal of immunopAralysis in pediatriC sEpsis-induced MODS Study
Acronym: GRACE
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Nationwide Children's Hospital (Other)
Responsible Party: Principal Investigator, Mark Hall, Professor, Department of Pediatrics, Nationwide Children's Hospital
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: GRACE
Record Dates: First submitted 2018-12-06; First posted 2018-12-10 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Pediatric Sepsis-induced MODS
Keywords: sepsis; MODS; pediatric; immunoparalysis; GM-CSF
MeSH Terms: conditions — Sepsis; Multiple Organ Failure | interventions — Granulocyte-Macrophage Colony-Stimulating Factor; Colony-Stimulating Factors; sargramostim

STUDY DESIGN:
Intervention Model Description: This is an open-label, sequential, dose- and route of administration-finding study that will be conducted in sequential cohorts of children with sepsis-induced MODS
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- IV GM-CSF 125 mcg/m2/dose (Experimental): Subjects in this arm who demonstrate immunoparalysis will receive GM-CSF by the intravenous (IV) route at a dose of 125 mcg/m2/day for 7 consecutive days.
  Interventions: Drug: GM-CSF
- SQ GM-CSF 125 mcg/m2/dose (Experimental): Subjects in this arm who demonstrate immunoparalysis will receive GM-CSF by the subcutaneous (SQ) route at a dose of 125 mcg/m2/day for 7 consecutive days.
  Interventions: Drug: GM-CSF
- IV GM-CSF 250 mcg/m2/dose (Experimental): If the IV 125 mcg/m2/dose arm is not successful in the first cohort of subjects, we will transition to 250 mcg/m2/day via the IV route for 7 consecutive days in a subsequent cohort.
  Interventions: Drug: GM-CSF
- SQ GM-CSF 250 mcg/m2/dose (Experimental): If the SQ 125 mcg/m2/dose arm is not successful in a cohort of subjects (or if the IV dose had to be escalated to 250 mcg/m2/dose), we will transition to 250 mcg/m2/day via the SQ route for 7 consecutive days in a subsequent cohort.
  Interventions: Drug: GM-CSF

INTERVENTIONS:
Drug: GM-CSF — Subjects demonstrating immunoparalysis (defined by a whole blood ex vivo LP-induced TNF-alpha production capacity < 200 pg/ml) will receive 7 days of GM-CSF treatment by either the IV or SQ route at a dose of either 125 or 250 mcg/m2/day for 7 days.
  Other Names: granulocyte macrophage colony-stimulating factor; Leukine

SUMMARY:
This study is an open-label, multi-center, interventional trial in which children with sepsis-induced MODS undergo surveillance immune function testing beginning on Day 2 of MODS. Those children who demonstrate immunoparalysis (TNF-alpha response <200 pg/ml) will receive a 7-day course of GM-CSF at a dose of 125 or 250 mcg/m2/day by either the intravenous (IV) or subcutaneous (SQ) route.

The goal of the study is to establish the dose and route of delivery that results in resolution of immunoparalysis (TNF-alpha response >=200 pg/ml) by the morning after the 3rd scheduled dose with persistent resolution of immunoparalysis on the morning after the 7th scheduled dose. Resolution of immunoparalysis in 8 out of the first 10 subjects in a study treatment arm represents a successful dose and route. The goal of this study will be achieved through the following Specific Aims:

Specific Aim 1. Establish the immunologic efficacy of GM-CSF administered by the IV and SQ routes in children with immunoparalysis in the setting of sepsis-induced MODS.

Specific Aim 2. Estimate the pharmacokinetic parameters by the IV and SQ GM-CSF administered in pediatric sepsis-induced MODS.

Specific Aim 3. Demonstrate the feasibility of screening, enrollment, drug delivery, and sample collection for a multi-center immunostimulation trial in children with sepsis-induced MODS.

ELIGIBILITY:
Inclusion Criteria:

* >= 40 weeks gestational age to <18 years; AND
* Onset of >=2 new organ dysfunctions (compared to pre-sepsis baseline) as measured by the Proulx criteria; AND
* Documented or suspected infection as the MODS inciting event.

Exclusion Criteria:

* Unable to collect a cumulative total of 20.5 mL of blood for this study due to research blood draw limits; OR
* Limitation of care order at the time of screening; OR
* Patients at high risk for brain death; OR
* Active (or planned within 7 days) immunosuppressive treatment for oncologic, transplant, or rheumatologic disease; OR
* Known primary immunodeficiency disorder; OR
* Diagnosis of myeloid leukemia, myelodysplasia, or autoimmune thrombocytopenia;OR
* Known allergy to GM-CSF; OR
* Documented hyperferritinemia (serum ferritin >= 500 ng/ml) during current sepsis event; OR
* Contraindication to SQ injection (ECMO); OR
* Burns where >5% of the total body surface area is affected; OR
* Renal replacement therapy at the time of screening; OR
* On ECMO or anticipated to require ECMO; OR
* Known pregnancy; OR
* Inability to collect and ship sample for immune testing on MODS Day 2; OR
* Previous enrollment in the GRACE study

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Estimated)
Dates: Start 2018-12-05 (Actual); Primary Completion 2023-12-05 (Estimated); Study Completion 2023-12-05 (Estimated)

PRIMARY OUTCOMES:
TNF-alpha response | Subjects will be screened for immunoparalysis throughout their first three weeks of sepsis-induced MODS
  Success in a cohort is defined as improvement in the whole blood ex vivo LPS-induced TNF-alpha production capacity (TNF response) to >= 200 pg/ml by the morning after the 3rd dose and persisting to the morning after the 7th dose in at least 8 out of 10 treated subjects within a cohort

CONTACTS AND LOCATIONS:
Overall Officials: Mark W Hall, MD, Principal Investigator — Nationwide Children's Hospital
Locations (8):
- United States (8):
  - UCLA Mattel Children's Hospital, Los Angeles, California
  - Benioff Children's Hospital/UCSF, San Francisco, California
  - Children's Hospital of Colorado, Aurora, Colorado
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Children's Hospital of Michigan, Detroit, Michigan
  - Nationwide Children's Hospital, Columbus, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
After subject enrollment and follow up have been completed, the DCC will prepare a final study database for analysis. A releasable database will be produced and completely de-identified in accordance with the definitions provided in the Health insurance Portability and Accountability Act (HIPAA). Namely, all identifiers specified in HIPAA will be recoded in a manner that will make it impossible to deduce or impute the specific identity of any patient. The database will not contain any institutional identifiers.
Supporting Information: CSR, Analytic Code
Time Frame: After subject enrollment and follow up have been completed. Data will be available indefinitely.
Access Criteria: The public use dataset will be available through the CPCCRN website